CLINICAL TRIAL: NCT02442999
Title: Sleep Apnea in Non-ovulating REI Patients: The SNORES Randomized Clinical Trial
Brief Title: The SNORES Randomized Clinical Trial
Acronym: SNORES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00020545
Record Dates: First submitted 2015-04-13; First posted 2015-05-13 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: PCOS; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Mass Screening; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Screen for Sleep Apnea (Experimental): Screen for sleep apnea, treat with continuous positive airway pressure (CPAP) if diagnosed with sleep apnea
  Interventions: Other: Screening for obstructive sleep apnea; Device: CPAP - continuous positive airway pressure

INTERVENTIONS:
Other: Screening for obstructive sleep apnea
  Arms: Screen for Sleep Apnea
Device: CPAP - continuous positive airway pressure
  Arms: Screen for Sleep Apnea

SUMMARY:
Randomized clinical trial among women with polycystic ovary syndrome (PCOS) who present for fertility treatment to evaluate the impact of screening for obstructive sleep apnea.

DETAILED DESCRIPTION:
The investigators' goal is to perform a randomized clinical trial among women with PCOS who present for infertility treatment. Our primary outcome is to determine if screening women with PCOS, and treating those with confirmed sleep apnea, will lead to more ovulatory cycles. Our sub-aims are to describe the rate of OSA and sleep symptoms in patients with PCOS, to see if current sleep questionnaires correlate to a diagnostic sleep study, to describe the correlation between OSA and biomarkers of glucose homeostasis in women with PCOS, to investigate health related quality of life between the groups, to compare perinatal outcomes between the groups, and to evaluate the composition of breastmilk among women who choose to breastfeed.

ELIGIBILITY:
Inclusion Criteria

* Females 18 - 50 years old.
* Receiving care from an Obstetrician / gynecologist or a Reproductive endocrinology infertility specialist
* Polycystic ovarian syndrome defined by the modified Rotterdam criteria
* Able to speak and understand as well as give informed consent in English

Exclusion Criteria

* Late onset congenital adrenal hyperplasia
* Cushings disease
* Androgen-secreting tumors
* Previous diagnosis of obstructive sleep apnea
* Current use of over the counter or prescribed sleep medications.

  * Examples of medications that exclude a patient from this study include but are not limited to Unisom, Ambien or Lunesta.
  * Patients who are taking non-prescribed herbal medications for sleep will not be excluded from the study. Examples of these include but are not limited to melatonin, chamomile, or valerian.
* Untreated thyroid disease
* Prolactin excess
* Patients with the following medical conditions will be excluded from the study as portable sleep apnea monitors are not indicated in patients with severe pulmonary disease, neuromuscular disease, or congestive heart failure.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Ovulatory cycles | 3 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - USF REI Lakeland, Lakeland, Florida
  - USF REI Sarasota, Sarasota, Florida
  - USF REI St. Petersburg, St. Petersburg, Florida
  - USF South Tampa Center, Tampa, Florida
  - USF Morsani, Tampa, Florida
  - USF REI Wesley Chapel, Wesley Chapel, Florida